CLINICAL TRIAL: NCT02078817
Title: Open-Label Intravenous Subanesthetic Ketamine for Adolescents With Treatment-Resistant Depression
Brief Title: Ketamine in Adolescents With Treatment-Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22225
Record Dates: First submitted 2014-02-27; First posted 2014-03-05 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Major Depressive Disorder
Keywords: Treatment-resistant
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ketamine (Experimental): Intravenous ketamine 0.5 mg/kg over 40 minutes will be given 6 times over 2 weeks.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — IV infusions of 0.5mg/kg of Ketamine hydrochloride over a 40-minute infusion period. Participants will receive a total of 6 doses over a 2-week period.

SUMMARY:
This study will test the use of ketamine for treatment of depression in adolescents that have not responded to other treatments. We will also examine neurobiological mechanisms of treatment.

DETAILED DESCRIPTION:
Depression frequently emerges during adolescence and is associated with severe outcomes. Current interventions do not lead to remission for many adolescents. Treatment-resistant depression (TRD) in adolescence is an ominous prognostic indicator for a lifetime of suffering and increased risk for suicide. Efforts should be directed toward novel interventions that could alter this perilous course. Theoretically, restoration of healthy development during this critical window would substantially improve outcomes over the lifespan.

Ketamine is a noncompetitive, high-affinity antagonist of the N-methyl-D-aspartate type glutamate receptor that has long been used for induction and maintenance of anesthesia in children and adults, and recently has been investigated for its rapid antidepressant effects. Randomized, double-blind, saline-controlled trials in adults with TRD have demonstrated that a single, subanesthetic infusion of intravenous (IV) ketamine at 0.5 mg/kg over 40 minutes can produce a rapid (within 2 hours) antidepressant response (Ibrahim et al., 2011; Zarate et al., 2006). Recent evidence suggests that serial doses of ketamine may be even more effective and may lead to more prolonged remission (aan het Rot et al., 2010; Murrough et al., 2012). Our current research at using serial dosing of IV ketamine among adult veterans with TRD over a 2-week period has shown promising results, with a response rate of 92% among the 12 participants to date.

No results from any studies examining effectiveness of either single-dose or serial-dose ketamine have yet been published in adolescents with TRD. Because of the ongoing neurodevelopment in adolescence, which is thought to confer enhanced neuroplasticity, it is possible that adolescents with TRD could show greater responses and more sustained remission than adults with TRD. The biological mechanisms of depression impacted by ketamine are only now being uncovered in adults (Zarate et al., 2013). Characterization of the neural mechanisms underlying ketamine response or non-response in adolescents with TRD will represent a significant advance. The specific aims of this preliminary study are as follows:

Aim #1: To determine the efficacy of repeated-dose subanesthetic IV ketamine among adolescent patients with TRD.

Hypothesis: Based on previous results in adults with TRD, we predict that response rates will improve over the course of six treatments of ketamine.

Aim #2: To explore durability of antidepressant response to repeated dose of IV ketamine in a 4-week observational period.

Hypothesis: Based on the inherent neuroplasticity in adolescence due to ongoing neurodevelopment, adolescents may show a more durable clinical response than has been seen in adults.

Aim #3: To study the neurobiological mechanisms of response to ketamine. We will examine relevant biological systems using several different brain imaging indices and measures of intracellular functioning from peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adolescents aged 12 to 18 years.
* Presence of recurrent major depression without psychotic features confirmed by the Kiddie-Schedule for Affective Disorders and Schizophrenia - Parent and Lifetime Version (Kaufman et al., 1997).
* Current depression severity measured by the Children's Depression Rating Scale (CDRS) (Poznanski, 1985) raw score greater than or equal to 36 at screening and the day ketamine is due to be received for the first time.
* Current depressive episode resistant to treatment, defined as failure to achieve remission (elimination of symptoms and restoration of pre-morbid psychosocial functioning) from at least 2 antidepressant trials of different pharmacological classes. Systematic evaluation of previous antidepressant trials will be assessed by using the Antidepressant Treatment History Form (Sackeim, 2001).
* If present, current antidepressant medication treatment must be dose stable for at least 2 months prior to beginning the study. (Patients will continue with current antidepressant treatment throughout the study. Based on our experience in current research at the VA Medical Center using serial ketamine for adult TRD, patients have shown positive results while continuing their current antidepressant treatment.)

Exclusion Criteria:

* Inability to speak English
* Inability or unwillingness to provide written informed consent
* A history of Mental Retardation or any Pervasive Developmental Disorder
* Current or lifetime diagnosis of schizophrenia, schizoaffective disorder, or psychosis Not Otherwise Specified.
* Family history with a first degree relative with schizophrenia, schizoaffective disorder, or psychosis Not Otherwise Specified.
* Diagnosis of seizures or other neurological disorders.
* Comorbid diagnosis of substance abuse or dependence, current or past.
* Clinically unstable medical illness.
* Current use of the following medications: any barbiturates, any narcotics, any non-benzodiazepine hypnotics at doses higher than zolpidem 10 mg qhs or equivalent for insomnia.
* For women: pregnancy (confirmed by baseline lab test).
* The presence of any MRI contra-indications such as MRI-incompatible metals in the body or claustrophobia.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2014-09; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Roy AV, Thai M, Klimes-Dougan B, Westlund Schreiner M, Mueller BA, Albott CS, Lim KO, Fiecas M, Tye SJ, Cullen KR. Brain entropy and neurotrophic molecular markers accompanying clinical improvement after ketamine: Preliminary evidence in adolescents with treatment-resistant depression. J Psychopharmacol. 2021 Feb;35(2):168-177. doi: 10.1177/0269881120928203. Epub 2020 Jul 9. PMID 32643995

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine
Started | 14
Completed | 13
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ketamine
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.9 (0.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Estimated intelligence quotient [Mean (Standard Deviation); unit: IQ] | 114.1 (56.96)
Socioeconomic Status (SES) [Mean (Standard Deviation); unit: units on a scale] — SES was measured using the Hollingshead Four Factor Index of Socioeconomic Status, an instrument measuring the marital status, retired/employed status, educational attainment, and occupational prestige of the parents of child participants. Parent education is rated on a 7-point scale. Parent occupation is coded on a 9-point scale. Education and occupation scores are then weighted to obtain a single score for each parent (range 8 to 66). For households with 2 parents, scores are averaged. Higher scores indicate greater socioeconomic status (more financial and social resources).
  units on a scale | 56.96 (7.45)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.7 (6)
Children's Depression Rating Scale-Revised Score [Mean (Standard Deviation); unit: units on a scale] — The CDRS-R measure is given in interview form to child and parent separately. A consensus is then created with best-estimate for 17 items (each with a range of 1-5 or 1-7) using both sources of information. The total score is the sum of 17 item scores, ranging from 17-113 with higher scores indicating greater depression symptoms.
  units on a scale | 63.9 (12)
Beck Depression Inventory-II [Mean (Standard Deviation); unit: units on a scale] — BDI-II is a 21-item self-report multiple-choice inventory that assesses the severity of depressive symptoms over the prior week. Items are rated on a 4-point scale ranging from 0 to 3. Total scores are a sum of the 21 item scores ranging from 0 to 63. Higher scores indicate more severe depression symptoms.
  units on a scale | 29 (10)
Montgomery-Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — MADRS is a 10-item clinician-administered inventory measuring depression symptoms. Items are scored on a scare from 0 (none) to 6 (constant). Total scores are a sum of the 10 item scores, ranging from 0 to 60, with higher scores indicating greater symptom severity.
  units on a scale | 30.15 (5)
Age of depression onset [Mean (Standard Deviation); unit: years] | 12.6 (2.9)
Duration of current depressive episode [Mean (Standard Deviation); unit: years] | 3.8 (1.6)
Number of Past Treatments [Mean (Standard Deviation); unit: Past treatments] | 5.7 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders Measured by Clinical Global Impression (CGI)
Description: Responders will be defined as those with CGI ratings (given by the study clinician) of 1 or 2 (much or very much improved). Patients that are given a scores of 3-7 (minimally improved to very much worse) will be considered non-responders.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine
Number analyzed (Participants) | 13
Participants | 5

2. Secondary Outcome: Children's Depression Rating Scale-Revised
Description: The CDRS-R measure is given in interview form to child and parent separately. A consensus is then created with best-estimate for 17 items (each with a range of 1-5 or 1-7) using both sources of information. The total score is the sum of 17 item scores, ranging from 17-113 with higher scores indicating greater depression symptoms.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 13
score on a scale | 44.1 (16.3)

3. Secondary Outcome: Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: MADRS is a 10-item clinician-administered inventory measuring depression symptoms. Items are scored on a scare from 0 (none) to 6 (constant). Total scores are a sum of the 10 item scores, ranging from 0 to 60, with higher scores indicating greater symptom severity.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 13
score on a scale | 18.5 (11.2)

4. Secondary Outcome: Beck Depression Inventory-II (BDI-II)
Description: BDI-II is a 21-item self-report multiple-choice inventory that assesses the severity of depressive symptoms over the prior week. Items are rated on a 4-point scale ranging from 0 to 3. Total scores are a sum of the 21 item scores ranging from 0 to 63. Higher scores indicate more severe depression symptoms.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 13
score on a scale | 17.8 (15.7)

5. Secondary Outcome: Change in Clinician Administered Dissociative States Scale (CADSS)
Description: CADSS is a 27-item instrument measuring symptoms of dissociative stress, with 19 items completed by the patient and 8 items completed by the clinician. Items are rated on a scale of 0 (not at all) to 4 (extreme). Total scores are a sum of the 27 item scores and range from 0 to 108, with higher scores indicating greater symptom severity.
Time Frame: baseline, 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 13
score on a scale | -19.8 (14.8)

6. Secondary Outcome: Maximum Change in Systolic Blood Pressure
Description: Vital signs were measured every 15 minutes, starting from the beginning of the infusion and ending 2 hours after the infusion ended (2 hours, 40 minutes total). Maximum increase of blood pressure compared to baseline was calculated.
Time Frame: 2 hours and 40 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ketamine
Number analyzed (Participants) | 13
mmHg | 13.9 (9.4)

7. Secondary Outcome: Maximum Change in Diastolic Blood Pressure
Time Frame: baseline, 45 minutes post infusion
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ketamine
Number analyzed (Participants) | 13
mmHg | 13.6 (11.7)

8. Secondary Outcome: Maximum Change in Heart Rate
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Ketamine
Number analyzed (Participants) | 13
beats per minute | 8.9 (8.8)

9. Secondary Outcome: Maximum Decrease in Pulse Oximetry
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Ketamine
Number analyzed (Participants) | 13
percent | -2.5 (9.4)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 5/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=13)
Nausea (Gastrointestinal disorders) | 3 (3)
Headache (General disorders) | 1 (1)
Hand Pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT02078817/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT02078817/Prot_SAP_001.pdf